CLINICAL TRIAL: NCT02131584
Title: Administration of Jakafi (Ruxolitinib) for Symptom Control of Patients With Chronic Lymphocytic Leukemia (CLL): A Phase II Study
Brief Title: Ruxolitinib Phosphate in Reducing Fatigue in Patients With Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-0044; NCI-2014-01465 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0044 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (ruxolitinib phosphate) (Experimental): Patients receive ruxolitinib phosphate PO BID (approximately 12 hours apart) for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Questionnaire Administration; Drug: Ruxolitinib Phosphate

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi

SUMMARY:
This phase II trial studies how well ruxolitinib phosphate works in reducing fatigue in patients with chronic lymphocytic leukemia. Ruxolitinib phosphate may stop the growth of cancer cells by blocking a protein called Janus kinase (JAK) that is needed for cell growth and may also help control fatigue, decrease the size of lymph nodes and/or lower the number of chronic lymphocytic leukemia cells in the blood.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the reduction in fatigue as measured by the Brief Fatigue Inventory (BFI) of patients with chronic lymphocytic leukemia (CLL) who do not require anti-neoplastic therapy according to the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 recommendations.

SECONDARY OBJECTIVE:

I. To estimate the reduction in other symptoms using the M. D. Anderson Symptom Inventory (MDASI) and to assess disease burden and response by the IWCLL 2008 response criteria.

OUTLINE:

Patients receive ruxolitinib phosphate orally (PO) twice daily (BID) (approximately 12 hours apart) for up to 2 years in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to understand and sign an informed consent document
* Subjects must be diagnosed with CLL and do not meet the IWCLL criteria for treatment
* Patients may have been previously treated or previously untreated
* Symptomatic patients with a BFI symptom scale of 2 points or greater
* Subjects with hemoglobin values at the screening visit equal to or greater than 12.0 g/dL
* Subjects with a platelet count of at least 75 x 10^9/L at the screening visit
* Subjects with an absolute neutrophil count (ANC) of equal to or higher than 0.5 x 10^9/L at the screening visit
* Subjects must have discontinued all drugs used to treat CLL no later than day -30
* Subjects with an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2

Exclusion Criteria:

* Females who are pregnant or are currently breastfeeding
* Subjects of childbearing potential who are unwilling to take appropriate precautions (throughout the study from screening, including 30 days after discontinuation of the study drug) to avoid becoming pregnant or fathering a child

  * Females of non-childbearing potential are defined as women who (a) are equal to or greater than 55 years of age with history of amenorrhea for 1 year, or (b) are surgically sterile for at least 3 months
  * For females of childbearing potential, or for males, appropriate precautions are those that are at least 99% effective in preventing the occurrence of pregnancy; these methods should be communicated to the subjects and their understanding confirmed:

    * Complete abstinence from sexual intercourse
    * Double barrier methods
    * Condom with spermicide in conjunction with use of an intrauterine device (IUD)
    * Condom with spermicide in conjunction with use of a diaphragm
    * Oral, injectable, or implanted contraceptives
    * Tubal ligation or vasectomy (surgical sterilization)
* Subjects with recent history of inadequate bone marrow reserve as demonstrated by previous transfusions except for acute blood loss (e.g. surgery) in the month prior to screening
* Alanine aminotransferase (ALT) > 2.5 x upper limit of normal (ULN)
* Modification of diet in renal disease (MDRD) calculated glomerular filtration rate (GFR) < 30 mL/min
* Subjects with active uncontrolled infection or who are human immunodeficiency virus (HIV) positive (subjects with acute infections requiring treatment should delay screening/enrollment until the course of therapy has been completed and the event is considered controlled)
* Subjects with an invasive malignancy over the previous 2 years except treated basal or squamous carcinomas of the skin completely resected intraepithelial carcinoma of the cervix and completely resected papillary thyroid and follicular thyroid cancers; other completely resected cancers greater than 2 years may be considered after review by the principal investigator (PI)
* Subjects with clinically significant uncontrolled cardiac disease
* Subjects being treated concurrently with any prohibited medications, including investigational medication, rifampin, St. John's wort, and potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors (excluding ketoconazole) unless continuation of such medications are determined by the investigator to be in the best interest of the patient
* Subjects who have previously received JAK inhibitor therapy
* Subjects with active alcohol or drug addiction that would interfere with their ability to comply with the study requirements
* Subjects with any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol
* Subjects who have unknown transfusion history for at least the 12 weeks prior to screening
* Subjects who are unable to complete the symptom diary
* Subjects who will need conventional therapy during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue | Baseline to 3 months
  As measured by the Brief Fatigue Inventory (BFI) question 3 regarding the worst fatigue in the past 24 hours. Will be analyzed in a continuous fashion.

SECONDARY OUTCOMES:
Proportion of patients with 2 point reductions in the BFI #3 score | Up to 3 months
  Proportion of patients at 3 months versus at enrollment tabulated.
20% improvement in symptoms | Up to 3 months
  As measured by the M. D. Anderson Symptom Inventory (MDASI).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jain P, Keating M, Renner S, Cleeland C, Xuelin H, Gonzalez GN, Harris D, Li P, Liu Z, Veletic I, Rozovski U, Jain N, Thompson P, Bose P, DiNardo C, Ferrajoli A, O'Brien S, Burger J, Wierda W, Verstovsek S, Kantarjian H, Estrov Z. Ruxolitinib for symptom control in patients with chronic lymphocytic leukaemia: a single-group, phase 2 trial. Lancet Haematol. 2017 Feb;4(2):e67-e74. doi: 10.1016/S2352-3026(16)30194-6. Epub 2017 Jan 12. PMID 28089238
- See also: M D Anderson Cancer Center — http://www.mdanderson.org